CLINICAL TRIAL: NCT07075796
Title: Study of the Performance of the GLUCUBE System in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iGluco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-NIGM-004
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: non-invasive glucose measurement; diabetes; tipo 2; glucometer
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-Label (Other): GLUCUBE system performance in the monitoring and measurement of the blood glucose compared to the standard glucometer (blood capillary glucometer - Bayer Contour®Next).
  Interventions: Device: GLUCUBE system

INTERVENTIONS:
Device: GLUCUBE system — A non-invasive system to monitor and measure the blood glucose compared to the standard glucometer in a group subjects

SUMMARY:
This study is a prospective, single center, open label clinical investigation. The primary objective of the study is to evaluate the performance of GLUCUBE in patients with diabetes type 2 and how the accuracy of the system improves as the time of use by the patient increases.

DETAILED DESCRIPTION:
Current methods of measuring blood glucose, glucometers, although minimally invasive, can be painful as they require puncturing the fingertip with a prick device and drawing a drop of blood, which is applied to a disposable test strip. This minimal invasiveness can cause discomfort and discourage the user from testing their blood glucose levels as frequently as necessary, leading to poor glycemic control. Due to the non-invasive nature of the GLUCUBE system, it provides glucose level information safely and painlessly, avoiding any discomfort to the user. It is low cost as it uses commonly used electronic components and does not require test strips or other consumables that would increase the ongoing cost of the device. The performance of the GLUCUBE system has already been evaluated in comparison to the standard glucometer (Ascensia Contour®Next) in adult patients with and without diabetes. The primary objective of this clinical investigation is to evaluate the performance of GLUCUBE in patients with diabetes type 2 and how the accuracy of the system improves as the time of use by the patient increases.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age.
* Diagnosed with type 2 diabetes mellitus.
* Have a smartphone with an internet connection that allows the installation of the GLUCUBE APP.
* Be able to use the GLUCUBE system autonomously, in the opinion of the researcher.
* Have signed the informed consent.

Exclusion Criteria:

* The patient is currently participating in another clinical investigation or has participated in another clinical investigation in the last 30 days prior to the start of this study.
* Pregnant or breast-feeding women and those subjects who plan pregnancy during the clinical investigation follow-up period.
* Presence of other anatomical or comorbid conditions, or other medical, social or psychological conditions that, in the opinion of the investigator, could limit the subject's ability to participate in the clinical investigation or to comply with the follow-up requirements, or affect the scientific soundness of the clinical investigation results.
* Patients with any active and/or infectious acute illness.
* Patients who have a condition that affects blood circulation in the fingers of the hand, such as Raynaud's phenomenon.
* Any medical condition that, in the opinion of the investigator, will increase the risk of hyperglycemic and hypoglycemic events: seizures, heart disease, unconscious hypoglycemia, etc.
* Patients with an inability to maintain hand stability during measurement or with progressive nervous system disease affecting movement (Parkinson's disease, moderate-severe essential tremor, and other diseases with involuntary movements).
* Patients suffering from calluses, malformations, or open wounds with bandages on their hands.
* Patients with nail polish or any type of false nail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Performance Evaluation | 4 times/day for 1 week
  Performance of the GLUCUBE device in monitoring and measuring blood glucose in adult patients with type 2 diabetes, compared to the standard glucometer (capillary blood glucometer - Ascensia Contour®Next).
Performance Improvement Evaluation | through study completion, an average of 21 days
  Improved performance of the GLUCUBE device as patient usage time increases.

OTHER OUTCOMES:
User Satisfaction | 21 days after the participant enters the study
  Evaluation of patient preferences for using the GLUCUBE system versus a capillary glucometer. Device(s) to be used in clinical research.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Especialidades Virgen de los Reyes. Hospital Universitario Virgen del Rocío, Seville, Seville, Spain